CLINICAL TRIAL: NCT00585689
Title: A Phase Two Trial of Neoadjuvant ABI-007, Carboplatin and Gemcitabine in Patients With Locally Advanced Carcinoma of the Bladder
Brief Title: Neoadjuvant ABI-007, Carboplatin and Gemcitabine in Locally Advanced Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.061; HUM 13486 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Bladder Cancer
Keywords: Locally advanced urothelial carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Albumin-Bound Paclitaxel; Carboplatin; Gemcitabine; Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant ABI-007, Carboplatin, and Gemcitabine (Experimental): Neoadjuvant ABI-007 (260 mg/m^2) on day 1, Carboplatin (Target AUC [Area under the curve] =5) on day 1, and Gemcitabine (800 mg^m2) on days 1 and 8, every 21 days.
  Interventions: Drug: ABI-007; Drug: Carboplatin; Drug: Gemcitabine; Procedure: Radical Cystectomy

INTERVENTIONS:
Drug: ABI-007 — ABI-007 will be administered at a dose of 260 mg/m2 over a 30 min IV infusion on day 1 of each 21 day cycle.
Drug: Carboplatin — Carboplatin will be administered at a dose of TARGET AUC=5 over a 15 min IV infusion of day 1 of each 21 day cycle.
Drug: Gemcitabine — Gemcitabine will be administered at a dose of 800 mg/m2 over a 30 min IV infusion on days 1 and 8 of each 21 day cycle.
Procedure: Radical Cystectomy

SUMMARY:
Study participants will have been diagnosed with bladder cancer that has invaded the muscle wall of the bladder. Surgery is used to remove cancer when it is in the muscle of the bladder. Unfortunately, approximately 50% of people may have their cancer return in another location. For this reason, researchers are focusing on new chemotherapy regimens to be given before surgery (to remove the bladder) that may decrease the likelihood of cancer spreading.

Paclitaxel, carboplatin and gemcitabine are chemotherapy drugs known to destroy bladder cancer cells.

ABI-007 (brand name Abraxane™) is a form of the chemotherapy drug called paclitaxel. Standard paclitaxel is formulated with ethanol and a substance called Cremophor EL (polyoxyethylated castor oil). However, these additives are felt to contribute to the side effects (possibly severe) associated with paclitaxel. ABI-007 does not contain these additives and may deliver more drug to tumor cells. ABI-007 is approved by the United States Food and Drug Administration (FDA) in the treatment of metastatic (advanced) breast cancer, and is being evaluated in other cancers in research studies.

This study will evaluate the safety and efficacy of the combination of ABI-007, carboplatin and gemcitabine in the treatment of bladder cancer prior to surgery to remove the bladder.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced (T2-4,N0,M0 or Tany,N1-3,M0) urothelial carcinoma of the bladder and be candidates for cystectomy following chemotherapy. Tumor specimens must be available for assay of molecular markers (correlative research).
* Performance status of 0, 1 or 2 by Eastern Cooperative Oncology Group (ECOG) criteria.
* Serum creatinine <2.0 mg/dl and/or creatinine clearance >40 ml/min.
* Granulocyte count > 1,500/mm3, platelet > 100,000/mm3, and hemoglobin > 9.0 g/dl.
* Adequate liver functions: AST and ALT < 2.5 X upper limit of normal, alkaline phosphatase < 2.5 X upper limit of normal, and bilirubin < 1.5 mg/dl.
* Pre-existing peripheral neuropathy > grade 2
* Recovered from any effects of surgery.
* Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Women with reproductive potential must have a negative pregnancy test.

Exclusion Criteria:

* Prior systemic or intra-arterial chemotherapy and rior radiotherapy. (intravesical chemotherapy allowed.)
* Pre-existing peripheral neuropathy > grade 2
* Prior malignancy [except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease free for 2 years]
* Unresolved bacterial infection requiring active treatment with antibiotics. (Treatment may begin at the conclusion of antibiotic therapy.)
* Pregnant or lactating women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Smith, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Grivas PD, Hussain M, Hafez K, Daignault-Newton S, Wood D, Lee CT, Weizer A, Montie JE, Hollenbeck B, Montgomery JS, Alva A, Smith DC. A phase II trial of neoadjuvant nab-paclitaxel, carboplatin, and gemcitabine (ACaG) in patients with locally advanced carcinoma of the bladder. Urology. 2013 Jul;82(1):111-7. doi: 10.1016/j.urology.2013.03.044. Epub 2013 May 21. PMID 23706253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine
Started | 29
Completed | 22
Not Completed | 7
Not completed — Received different ABI-007 schedule | 3
Not completed — Adverse Event | 1
Not completed — Patient Declined Surgery | 1
Not completed — Patient had unresectable disease | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 66 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Performance Status (ECOG) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is an attempt to quantify cancer patients' general well-being and activities of daily life. The score runs from 0 to 5, with 0 denoting perfect health and 5 death.
  participants
    0 | 17
    1 | 12
Clinical Disease Stage [Number; unit: participants]
  T2N0 | 18
  T2N1 | 2
  T2N2 | 1
  T3N0 | 6
  T4N0 | 2
Hydronephrosis Present [Number; unit: participants]
  Yes | 8
  No | 21
Angiolymphatic Invasion Present [Number; unit: participants]
  Yes | 9
  No | 20
Adjacent Carcinoma in Situ Present [Number; unit: participants]
  Yes | 16
  No | 13
Mixed Histological Features Present [Number; unit: participants]
  70% Plasmacytoid, 5% Sarcomatoid | 1
  10% Plasmacytoid, 10% Signet Ring | 1
  5% Squamous | 1
  10% Spindle | 1
  20% Glandular | 1
  Nested | 3
  Micropapillary | 1
  Micropapillary and Nested | 1
  None | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Pathologic Response After 3 Cycles of Treatment
Description: The rate of pathologic complete response (pT0) following three 21 day cycles of neoadjuvant ABI-007, carboplatin and gemcitabine was determined.
Time Frame: 63 days (post 3 cycles)
Population: 29 patients were enrolled. 26 of the 29 patients received the planned 3 cycles. 22 of the 26 patients had a cystectomy and were evaluable for the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine
Number analyzed (Participants) | 22
percentage of patients | 27.3 [10.7 to 50.2]

ADVERSE EVENTS:
Arm/Group | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine
Serious Adverse Events (participants affected / at risk) | 26/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine (N=29)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 22 (34)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Flu-like syndrome (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant ABI-007, Carboplatin, and Gemcitabine (N=29)
Anemia (Blood and lymphatic system disorders) | 19 (32)
Leukopenia (Blood and lymphatic system disorders) | 19 (37)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 25 (59)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (46)
Hypertension (Cardiac disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 25 (32)
Rigors/chills (General disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 22 (25)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 (6)
Hot flashes/flushes (Vascular disorders) | 3 (3)
Anorexia (Gastrointestinal disorders) | 11 (11)
Constipation (Gastrointestinal disorders) | 8 (9)
Dehydration (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 15 (18)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (5)
Febrile neutropenia (Infections and infestations) | 4 (4)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 2 (2)
Edema: limb (General disorders) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (8)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (6)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (10)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 3 (3)
Neuropathy: sensory (Nervous system disorders) | 17 (20)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Limb Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Headache Pain (Nervous system disorders) | 3 (3)
Joint Pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Pelvic Pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Pain - Other (Specify) (General disorders) | 4 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cystitis (Renal and urinary disorders) | 3 (3)
Urinary frequency/urgency (Renal and urinary disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes